CLINICAL TRIAL: NCT00303511
Title: Pacemaker Therapy in Adults With Congenital Heart Defects
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Wendy M. Book, Principal Investigator, Emory University
Other Study IDs: 0103-2006
Record Dates: First submitted 2006-03-16; First posted 2006-03-17 (Estimated); Results first posted 2014-08-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-07

CONDITIONS: Congenital Disorder
Keywords: adult; pacemaker; bradycardia; tachycardia; heart failure
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Bradycardia; Tachycardia; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Review the feasibility, safety and outcomes in adults with congenital heart disease who undergo pacemaker implantation for bradycardia, tachycardia or heart failure indications

DETAILED DESCRIPTION:
Survival to adulthood is now common for children born with congenital heart defects (CHD). This improved survival is in large part due to advances in cardiac surgery over the past 4 decades. However, few cardiac surgical repairs are curative. Many 'repaired' children with congenital heart defects later develop problems as adults. Arrhythmias, need for additional surgery, and heart failure are the more common late sequelae of congenital heart disease (1). In addition, many adults with CHD will need a pacemaker for sick sinus syndrome (inability of the inherent pacemaker of the heart to function properly resulting in bradycardia sometimes alternating with tachycardia), tachyarrhythmias or heart block (2, 3). Certain group of patients, such as those with congenital corrected transposition of the great arteries (CCTGA), d-transposition s/p atrial switch procedures and those with single ventricle physiology are at particular risk of developing heart failure (4). Attached figures show the anatomy of these congenital heart defect. Cardiac resynchronization therapy improves exercise tolerance, symptoms and reduces mortality in adults with heart failure due to acquired left ventricular dysfunction.(5-8). In addition, automatic internal cardioverter - defibrillators (ICD) have now been shown to decrease mortality in patients with low ejection fraction due to ischemic or non-ischemic etiologies (9, 10).

Patients with CHD pose a challenge to traditional transvenous pacemaker lead placement due to either complex venous anatomy that precludes conventional percutaneous approaches for pacemaker implantation or occlusions of central venous form multiple prior procedures (11, 12). As evident in the study by Janousek et.al, 7 out of 8 patients enrolled in this study required a thoracotomy for lead placement (4). While thoracoscopic epicardial lead placement has been described for placement of pacemaker leads in adults without congenital heart defects (13, 14), it has not been described for adult patients with congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Congenital heart disease diagnosis
* Pacemaker implantation completed during the period of Jan. 1, 1996 to Dec. 1, 2005
* Age 18 to 80, inclusive

Exclusion Criteria:

* Those who do not meet inclusion criteria

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with congenital heart disease requiring epicardial pacemaker leads
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 1996-01; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy M Book, MD, Principal Investigator — Emory University SOM
Locations (1):
- Emory University SOM Adult Cardiac Clinic, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: retrospective chart review
Period: Overall Study
Arm/Group | ACHD With Pacemaker
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ACHD With Pacemaker
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Pacemaker Implant With Total Thoracoscopic Approach to Epicardial Pacing Lead
Description: The ability to place a pacemaker with capture (have the pacemaker work properly) through totally thoracoscopic approach to epicardial pacing lead without requiring conversion to open procedure
Time Frame: 30 days
Measure: Number; unit: percentage of particiapants
Arm/Group | Cohort
Number analyzed (Participants) | 10
percentage of particiapants | 100

ADVERSE EVENTS:
Time Frame: retrospective study
Description: retrospective study, observational, not interventional
Arm/Group | ACHD With Pacemaker
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes